CLINICAL TRIAL: NCT06627374
Title: The Predictive Value of Thoracic Ultrasound As a Response to the Closure of Hemodynamically Significant Patent Ductus Arteriosus in Premature Infants: an Observational Pilot Study
Brief Title: Study of Thoracic Ultrasound As a Response to the Closure of Hemodynamically Significant Patent Ductus Arteriosus in Premature Infants
Acronym: LUNG PDA
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Paladini Angela, Consultant, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6973
Record Dates: First submitted 2024-09-26; First posted 2024-10-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Patency of the Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Patent Ductus Arteriosus in neonates — Neonates admitted to Neonatal care Unit after birth, undergoing hsPDA (hemodynamically significant Patent Ductus Arteriosus) closure according to standard clinical practice, will be included.

SUMMARY:
The diagnostic hypothesis is based on the evidence that, while the functional closure of the PDA (Patent Ductus Arteriosus) occurs within a few hours after birth, anatomical closure may take several weeks. The functional closure of the PDA can be extremely sensitive to variations in blood oxygen tension and the hemodynamic instability of preterm infants. Therefore, echocardiographic evaluation and ductal diameter at a single point in time (such as during PDA echocardiography) may not correlate with transductal blood flow. Assessing the variation in the amount of pulmonary interstitial fluid using LUS (lung ultrasound score) could be an early predictive parameter for the closure or non-closure of hsPDA (hemodynamically significant PDA).

ELIGIBILITY:
Inclusion Criteria:

* Neonates under 28 days of life
* Patients eligible for hsPDA closure treatment according to standard clinical practice

Exclusion Criteria:

* Neonates with congenital heart diseases (except for PDA and patent foramen ovale)
* Neonates with pneumothorax
* Neonates with pulmonary hemorrhage

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Full-term and preterm neonates admitted to the aforementioned operational unit after birth, undergoing closure of the hsPDA (hemodynamically significant Patent Ductus Arteriosus) according to standard clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Lung ultrasound score variability | From enrollment to the end of treatment on average of 3 - 15 days
  To assess the changes, particularly any reduction in the lung ultrasound score (LUS), during the closure of the hemodynamically significant PDA, according to standard clinical practice. The LUS score can range from 0 to 12. Higher values correspond to a greater overflow of fluids in the lungs.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, roma, Italy

IPD SHARING:
Plan to Share IPD: No